CLINICAL TRIAL: NCT02029599
Title: A Phase 2 Randomised, Double-blind, Placebo-controlled Multiple Ascending Dose Study Evaluate the Efficacy and Safety of Fang yi Qing Feng Shi Granules in Subjects With Rheumatoid Arthritis
Brief Title: The Efficacy and Safety of Fang yi Qing Feng Shi Granules in Subjects With Rheumatoid Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Maoxiang Group Jilin Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: China.JLMXFYQ2008-01
Record Dates: First submitted 2013-12-26; First posted 2014-01-08 (Estimated); Last update posted 2015-10-09 (Estimated); Status verified 2015-10

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Methotrexate; Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- High dose group (Experimental): Fang yi qing feng shi granule, Oral,10g, 3 times a day, Oral,for 3 months Methotrexate,Oral,7.5-15mg per week Acetaminophen tablets,Oral,0.5g, 1~2 times a day, when vas=10.
  Interventions: Drug: Fang yi qing feng shi granule; Drug: Methotrexate; Drug: Acetaminophen tablets
- Low dose group (Experimental): Fang yi qing feng shi granule,Oral,10g, 2 time a day, taking morning and evening,for 3 months.
  placebo,Oral,10g, 1 time a day, taking noon ,for 3 months. Methotrexate,Oral,7.5-15mg per week. Acetaminophen tablets,Oral,0.5g, 1~2 times a day, when vas=10.
  Interventions: Drug: Fang yi qing feng shi granule; Drug: placebo; Drug: Methotrexate; Drug: Acetaminophen tablets
- The placebo group (Placebo Comparator): placebo,Oral,10g, 3 time a day ,for 3 months. Methotrexate,Oral,7.5-15mg per week. Acetaminophen tablets,Oral,0.5g, 1~2 times a day, when vas=10.
  Interventions: Drug: placebo; Drug: Methotrexate; Drug: Acetaminophen tablets

INTERVENTIONS:
Drug: Fang yi qing feng shi granule — 10g, Oral,Three each time, 3 times a day,for 3 months;
  Arms: High dose group; Low dose group
Drug: placebo — 10g, Oral,Three each time, 3 times a day,for 3 months
  Arms: Low dose group; The placebo group
Drug: Methotrexate — 7.5-15mg per week，All patients should be used
Drug: Acetaminophen tablets — Oral,0.5g, 1~2 times a day, when vas=10

SUMMARY:
The aim of this study is to evaluate the efficacy and safety of Fang yi qing Feng shi granules in subjects with Rheumatoid Arthritis.

DETAILED DESCRIPTION:
Fang yi qing feng shi granules is the chinese patent medicine, which contains 8 kinds of chinese medicine .

Fang yi qing feng shi granules was approved by China Food and Drug Administration (CFDA) in 2005, produced by means of modern technology by Maoxiang Group Jilin Pharmaceutical Co., Ltd.The study is a multi-center, double -blind, placebo -controlled, randomized in Chinese subjects with Rheumatoid Arthritis to assess treatment effect and safety in the subjects treated with Fang yi qing feng shi granules versus subjects treated with placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects have the diagnosis of Rheumatoid Arthritis in active state.
2. Subjects have the Traditional Chinese Medicine (TCM) diagnosis ofArthralgic Syndrome with the sign of dampness obstructing connecting vessel。
3. Subjects must stop the medicine at least three month，which is Diseases modifying anti-rheumatic drugs(including glucocorticoids).
4. Male or female subjects, between the ages of 18 and 65 years old.
5. Joint function grading and ray classification are both in Ⅰ～Ⅲ.
6. Subjects agree to participate in this study and sign the informed consent form.

Exclusion Criteria:

1. Subjects with systemic lupus erythematosus,sicca syndrome, or severe osteoarthropathy will be excluded.
2. Subjects with severe rheumatic arthritis are loss of ability
3. Allergic to test drugs(basic treatment or drug combination),Allergic constitution(Allergic to two or more drugs).
4. Female subject who was pregnant or breast-feeding or considering becoming pregnant.
5. Subjects with sever diseases in Cardiovascular, brain, lung, liver, kidney and hematopoietic system.
6. The Liver function (ALT,AST) and kidney function（BUN,Cr）is higher than normal.
7. The Blood Routine (leukocyte count,platelet count)is lower than normal.
8. Subject considered by the investigator, for any reason, to be an unsuitable candidate for the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2014-03; Primary Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
The percentage of Therapeutic effect with American College of Rheumatology standards (ACR) | Taken at day 1 (baseline) and Change from Baseline in 4th,8th,12th week

SECONDARY OUTCOMES:
The change of Rheumatoid Arthritis (RA) associated symptoms and signs | Taken at day 1 (baseline) and Change from Baseline in 4th,8th,12th week
  The symptoms and signs include "Tender joint count,swollen joint count,time of morning stiffness,mean grip strength, VAS score,Jint function"
Safety assessments will be based on adverse event reports and the results of vital sign measurements, electrocardiogram, physical examinations, and clinical laboratory tests | Taken at day 1 (baseline) and Change from Baseline in 4th,8th,12th week
The subjects of their comprehensive evaluation of disease activity(AIMS),The observer to the comprehensive evaluation of disease activity in the study(AIMS),The subjects of physical function evaluation(HAQ). | Taken at day 1 (baseline) and Change from Baseline in 4th,8th,12th week
The change of laboratory test indexes (ESR、RF、CRP) | baseline,week12
Traditional Chinese Medicine(TCM) characteristics evaluative index: Traditional Chinese medicine Syndrome Scale | Taken at day 1 (baseline) and Change from Baseline in 4th,8th,12th week
The score of clinical symptoms and symptom integral | Taken at day 1 (baseline) and Change from Baseline in 4th,8th,12th week
Change in the days and doses using of analgesic(Paracetamol Tablets) | Taken at day 1 (baseline) and Change from Baseline in 4th,8th,12th week

CONTACTS AND LOCATIONS:
Overall Officials: wei liu, Principal Investigator — First Teaching Hospital of Tianjin University of Traditional Chinese Medicine
Locations (5):
- China (5):
  - Hubei provincial hospital of tcm, Wuhan, Hubei
  - Hospital of Liaoning University of Traditional Chinese Medicine, Shenyang, Liaoning
  - LONGHUA Hospital Shanghai University of TCM, Shanghai, Shanghai Municipality
  - First Teaching hospital of Tianjin University of Traditional Chinese Medicine, Tianjin, Tianjin Municipality
  - Second affiliated hospital of Tianjin university of tcm, Tianjin, Tianjin Municipality